CLINICAL TRIAL: NCT00001209
Title: A Pilot Study for the Treatment of Patients With Metastatic and High Risk Sarcomas and Primitive Neuroectodermal Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 860169; 86-C-0169
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-09

CONDITIONS: Neuroectodermal Tumor, Primitive; Neuroepithelioma; Osteosarcoma; Sarcoma; Sarcoma, Ewing's
Keywords: Combined Chemotherapy; Irradiation; Unresectable
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive; Neuroectodermal Tumors; Osteosarcoma; Sarcoma; Sarcoma, Ewing | interventions — Vincristine; Doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: vincristine, adriamycin and cytoxan, alternating with ifosfamide VP-16

SUMMARY:
This protocol is designed to test the feasibility of the administration of vincristine, adriamycin and cytoxan, alternating with the newly developed regimen ifosfamide VP-16 as well as the efficacy of this therapy in addition to radiotherapy in producing complete responses and disease-free survival in patients with Ewing's sarcoma, primitive sarcoma of bone, peripheral neuroepithelioma, and soft tissue sarcoma. This will not be a randomized study but will be comparable to the large data base of similar patients treated on successive Pediatric Branch studies.

DETAILED DESCRIPTION:
This protocol is designed to test the feasibility of the administration of vincristine, adriamycin and cytoxan, alternating with the newly developed regimen ifosfamide VP-16 as well as the efficacy of this therapy in addition to radiotherapy in producing complete responses and disease-free survival in patients with Ewing's sarcoma, primitive sarcoma of bone, peripheral neuroepithelioma, and soft tissue sarcoma. This will not be a randomized study but will be comparable to the large data base of similar patients treated on successive Pediatric Branch studies.

ELIGIBILITY:
Patients with high grade soft tissue sarcomas and either metastatic disease or stage III tumors including synovial sarcoma, malignant fibrous histiocytoma, hemangiopericytoma, malignant schwannoma (neurofibrosarcoma).

Patients must not have been previously treated with chemotherapy or radiation therapy.

The patients age must be less than or equal to 25 years.

The patient (or their guardian if under 18 years of age) must sign a document indicating that he/she is aware of the investigational nature of this treatment protocol and the potential risks and benefits that may be expected.

Patients must have a direct bilirubin of less than 4.0 mg/dl.

Patients must not have abnormal cardiac function (ejection fraction greater than 45% on MUGA scan with confirmation of shortening-fraction greater than 25% on echocardiography).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1986-10; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States